CLINICAL TRIAL: NCT02256852
Title: Open Label,Single Arm,Exploratory Study to Evaluate the Safety,Tolerability,Compliance and MOA,of QBKPN SSI in Subjects With 2 or More Second Primary Pre-invasive/Invasive Adenocarcinoma Following Surgical Resection of Stage I NSCLC
Brief Title: Exploratory Study of QBKPN SSI in Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Qu Biologics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QBKPN-01
Record Dates: First submitted 2014-09-30; First posted 2014-10-06 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- QBKPN SSI (Experimental): Individualized maintenance dose administered subcutaneously for 12 weeks
  Interventions: Biological: QBKPN SSI

INTERVENTIONS:
Biological: QBKPN SSI — QBKPN SSI is administered subcutaneously for 12 weeks

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, compliance and mechanism of action of study drug (QBKPN SSI) in subjects with two or more second primary pre-invasive or invasive adenocarcinoma following surgical section of Stage 1 NSCLC.

DETAILED DESCRIPTION:
Please refer to summary above.

ELIGIBILITY:
Inclusion Criteria:

* Male or female who is at or above the age of consent
* Histologically confirmed original diagnosis of lung cancer
* Life expectancy greater than 12 months
* ECOG performance status 0, 1, or 2 at screening
* Female subjects who agree to practice two effective methods of contraception from the time of signing the informed consent form through one month after the last dose of study drug
* Male subjects who agree to practice effective barrier contraception during the entire study drug period and through one month after the last dose of study drug

Exclusion Criteria:

* Extra-thoracic lung cancer progression
* Any active malignancies
* Any uncontrolled or major organ dysfunction
* Any past or current radiation or systemic therapies for the treatment of lung cancer
* Known HIV infection or other immunosuppressive disorder
* Concurrently participating in another study with an investigational immunotherapy or have received investigational immunotherapy within 3 months prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-12; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Safety, tolerability and compliance variables | 16 weeks
  Assess the number of adverse events and subject reported data

SECONDARY OUTCOMES:
Exploratory variables | 16 weeks
  Assess and identify biomarkers associated with immune response

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Stephen Lam, Principal Investigator — British Columbia Cancer Agency
Locations (1):
- BC Cancer Research Centre, Vancouver, Canada